CLINICAL TRIAL: NCT06664073
Title: The Predictive Value of the HEARTRISK6 Scale in Predicting Short-Term Serious Outcomes in Emergency Department Acute Heart Failure Patients
Brief Title: Heart Risk 6 Scale in Emergency Department Acute Heart Failure Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Basma Mahrous Mohamed, Resident physician, Assiut University
Other Study IDs: Heart Risk 6 scale in HF
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Acute Heart Failure (AHF)
Keywords: Heart risk 6 scale; Acute heart failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients will be assessed by supervised cardiology residents in emergency department, within 24 hou: Patients will be assessed for standardized clinical variables by supervised cardiology residents in emergency department, within 24 hours from ED treatment.
  •Routine laboratory values will be collected, cardiac troponins and ECG.

SUMMARY:
Detect the predictive value of the HEARTRISK6 Scale in Predicting Short-Term Serious Outcomes in emergency department acute heart failure patients in Egyptian population

DETAILED DESCRIPTION:
Recently, the heartrisk6 scale was introduced to predict the short-term serious outcomes in emergency department acute heart failure patients. It was created from 3 cohorts from American and Canadian population. Since the Egyptian population differ from the American and Canadian population regarding the age at presentation with cardiovascular disease, risk factors and etiology of the acute heart failure, we sought to detect the applicability of this score on our population.

ELIGIBILITY:
Inclusion Criteria:

* patients who have appropriate symptoms (short-ness of breath or fatigue)(<7 days duration); with clinical signs of ﬂuid retention (pulmonary or peripheral) in the presence of an underlying abnormality of cardiac structure or function.

  * If in doubt, a beneﬁcial response to treatment (eg, a brisk diuresis accompanied by improvement in breathlessness) will be considered.

Exclusion Criteria:

* Patients who did not ﬁt the deﬁnition of AHF or who were clearly too ill to be considered for discharge after 24 hours from ED:

  * 1) resting oxygen saturation <85% on room air
  * 2) heart rate >120 beats/min;
  * 3) systolic blood pressure <85 mm Hg;
  * 4) confusion, disorientation, dementia;
  * 5) primary presentation for ischemic chest pain requiring treatment or with acute ischemic ST-Tchanges on initial electrocardiogram (ECG);

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute heart failure
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2024-10-27 (Estimated); Primary Completion 2025-10-27 (Estimated); Study Completion 2027-10-27 (Estimated)

PRIMARY OUTCOMES:
Detect the predictive value of the heart risk 6 scale | 1 month
  -Detect the predictive value of the HEARTRISK6 Scale in Predicting Short-Term Serious Outcomes in the emergency department acute heart failure patients.

SECONDARY OUTCOMES:
Describe the management and outcomes of ED patients with acute heart failure | 1
  -Describe the management and outcomes of ED patients with acute heart failure, identify the various etiologies of this presentation, and characteristics and risk factors of this population.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stiell IG, Clement CM, Brison RJ, Rowe BH, Borgundvaag B, Aaron SD, Lang E, Calder LA, Perry JJ, Forster AJ, Wells GA. A risk scoring system to identify emergency department patients with heart failure at high risk for serious adverse events. Acad Emerg Med. 2013 Jan;20(1):17-26. doi: 10.1111/acem.12056. PMID 23570474
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Stiell IG, Perry JJ, Eagles D, Yadav K, Clement CM, McRae AD, Yan JW, Mielniczuk L, Rowe BH, Borgundvaag B, Dreyer J, Brown EL, Nemnom MJ, Taljaard M. The HEARTRISK6 Scale: Predicting Short-Term Serious Outcomes in Emergency Department Acute Heart Failure Patients. JACC Adv. 2024 May 24;3(7):100988. doi: 10.1016/j.jacadv.2024.100988. eCollection 2024 Jul. PMID 39129980